CLINICAL TRIAL: NCT00208052
Title: Behavioral Indicators of Pain:Tool Development With Concurrent and Construct Validity
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Organization: Cincinnati VA Medical Center (U.S. Federal Agency)
Other Study IDs: 02-11-1-1EE
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purpose of the pilot study is to validate an assesment tool to be used in the assessment of pain in the verbal, congitively intact patient. The ultimate goal is to be able to validate this tool in the non-verbal/cognitively impaired patient.

DETAILED DESCRIPTION:
Patinets will be observed for 2 six hour periods. Patients will be videotaped; every 10 minutes: EMG reading will be obtained; hourly - vital signs, pain score and saliva cortisol from "spit" will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* In-patients with Pain diagnosis

Exclusion Criteria:

* Unable to talk and or understand basic instructions
* Under age 18 or over age 75
* Receiving pain medications regularly

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2004-01; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Veronica B Steffen, MSN,RN, Principal Investigator — VA Medical Center; Amy Pettigrew, PHD,RN, Principal Investigator — University of Cincinnati, College of Nursing and Health
Locations (1):
- VA Medical Center, Cincinnati, Ohio, United States